CLINICAL TRIAL: NCT06945250
Title: A Multimedia Presentation to Augment the Informed Consent Process for Anesthesia for Patients Undergoing Scheduled Caesarian Delivery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Eleanor Kenny, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00222960
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Caesarean Section
Keywords: Pregnancy; Cesarean Section; Consent Process; Surgical Procedure

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Intervention Group: Participants randomized to the intervention group will receive a link to the audiovisual presentation via e-mail to review prior to coming into the hospital for caesarean section.
  Interventions: Other: Experimental Audio Visual
- Control Group (No Intervention): Control Group: Participants randomized to the control group will not receive the link to the audiovisual presentation

INTERVENTIONS:
Other: Experimental Audio Visual — Participants in this group will receive the audiovisual presentation
  Arms: Intervention Group

SUMMARY:
The informed consent process is an important part of any surgical and anesthetic intervention. It is also perhaps the most intellectually demanding portion of interacting with the healthcare system for patients. Competent patients have full autonomy over which treatments they receive, and making an informed choice about the decision to undergo a treatment requires at minimum a discussion of the proposed intervention, its risks and benefits, and alternatives to the proposed intervention.

The objective is to improve the anesthesia informed consent process for patients undergoing elective Caesarean delivery through the use of a pre-recorded audiovisual presentation that discusses the logistical aspects of perioperative care and the risks and benefits of anesthesia which is provided to patients prior to meeting their anesthesiologist.

The hypothesis is that the use of an audiovisual presentation which explains the purpose and nature of anesthesia for Caesarean delivery provided to the patient at least 24 hours prior to their procedure will result in a 10% increase in the effectiveness of risk communication and treatment decision making as measured by the Combined Outcome Measure for Risk Communication and Treatment Decision Making Effectiveness (COMRADE) tool.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or over on the day of the procedure
2. Able to provide verbal and written informed consent for participation in the study
3. Primarily English-speaking patients (the audiovisual presentation will be available only in English

Exclusion Criteria:

1. Refusal or inability to participate or provide informed consent
2. Primarily non-English speaking patients
3. At the discretion of the attending anesthesiologist of record due to medical complexity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant females only
Enrollment: 70 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
COMRADE survey score | 1 Day after delivery of baby
  COMRADE score for risk communication and treatment decision making on a 100-point scale, ranging from 0 (decision-making not informed at all (poor)) to 100 (most informed decision possible (good))

SECONDARY OUTCOMES:
Demographic factors associated with increase in informed decision-making | 1 Day after delivery of baby
  Demographic factors associated with increase in informed decision-making including age, education level, history of prior Caesarean delivery, history of other anesthetics (such as labor epidurals or general anesthetics)
Level of subjective anxiety associated with the proposed anesthetic | 1 Day after delivery of baby
  Level of subjective anxiety associated with the proposed anesthetic based on a scale of 1-5 (1) strongly disagree, (2) disagree, (3) neither agree nor disagree, (4) agree, (5) strongly agree).
Level of subjective fear associated with the proposed anesthetic | 1 Day after delivery of baby
  Level of subjective fear associated with the proposed anesthetic measured on a scale of 1-5 (1) strongly disagree, (2) disagree, (3) neither agree nor disagree, (4) agree, (5) strongly agree)
Level of satisfaction with the anesthetic informed consent process | 1 Day after delivery
  Level of satisfaction with the anesthetic informed consent process based on a scale of 1-5 (1) strongly disagree, (2) disagree, (3) neither agree nor disagree, (4) agree, (5) strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Kenny, MD, Principal Investigator — Northwestern Univesity
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edwards A, Elwyn G, Hood K, Robling M, Atwell C, Holmes-Rovner M, Kinnersley P, Houston H, Russell I. The development of COMRADE--a patient-based outcome measure to evaluate the effectiveness of risk communication and treatment decision making in consultations. Patient Educ Couns. 2003 Jul;50(3):311-22. doi: 10.1016/s0738-3991(03)00055-7. PMID 12900105
- [Background] Cassady JF Jr, Wysocki TT, Miller KM, Cancel DD, Izenberg N. Use of a preanesthetic video for facilitation of parental education and anxiolysis before pediatric ambulatory surgery. Anesth Analg. 1999 Feb;88(2):246-50. doi: 10.1097/00000539-199902000-00004. PMID 9972735
- [Background] Wisselo TL, Stuart C, Muris P. Providing parents with information before anaesthesia: what do they really want to know? Paediatr Anaesth. 2004 Apr;14(4):299-307. doi: 10.1046/j.1460-9592.2003.01222.x. PMID 15078374
- [Background] Atsaidis Z, Antel R, Guadagno E, Wiseman J, Poenaru D. Understanding the effectiveness of consent processes and conversations in pediatric surgery: A systematic-scoping review. J Pediatr Surg. 2022 Dec;57(12):834-844. doi: 10.1016/j.jpedsurg.2022.08.004. Epub 2022 Aug 11. PMID 36031429
- [Background] Garden AL, Merry AF, Holland RL, Petrie KJ. Anaesthesia information--what patients want to know. Anaesth Intensive Care. 1996 Oct;24(5):594-8. doi: 10.1177/0310057X9602400516. PMID 8909673
- [Background] Jawaid M, Farhan M, Masood Z, Husnain S. Preoperative informed consent: is it truly informed? Iran J Public Health. 2012;41(9):25-30. Epub 2012 Sep 1. PMID 23193502
- [Background] Tait AR, Teig MK, Voepel-Lewis T. Informed consent for anesthesia: a review of practice and strategies for optimizing the consent process. Can J Anaesth. 2014 Sep;61(9):832-42. doi: 10.1007/s12630-014-0188-8. Epub 2014 Jun 5. PMID 24898765